CLINICAL TRIAL: NCT02255331
Title: The Ability Of MRI To Detect Adverse Local Tissue Reaction And Implant Integration As A Function Of Hip Implant Modularity
Brief Title: Using MRI To Detect Soft Tissue Reactions And Implant Integration As Related To Implant Modularity
Status: Recruiting | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-442 R01 AR064840
Record Dates: First submitted 2014-08-28; First posted 2014-10-02 (Estimated); Last update posted 2025-06-19 (Actual); Status verified 2024-06

CONDITIONS: Complications; Arthroplasty; Complications; Arthroplasty, Mechanical
Keywords: Arthroplasty; Replacement; Hip; MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. A small sample of soft tissues surrounding a total hip replacement will be retained for histological evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrieval Analysis: You qualify for this Retrieval Analysis study if you:
  1. Have a total hip replacement with a ceramic component undergoing revision for any reason, including recurrent dislocation.
  2. Have a metal-on-polyethylene total hip replacement and have repeated dislocation, or
  3. Have a metal-on-polyethylene total hip replacement greater than 1 year old, or
  4. Have an infected total hip replacement (any surface bearing)
  You do not qualify for this arm of the study if you:
  1. Have occupational exposure to cobalt or chromium
  2. Presence of a metal-on-metal (MOM) implant, or a recalled implant
  3. Have had a prior revision of your total hip
  4. Standard contra-indications to MRI (e.g. cardiac pacemaker, etc.)
- Longitudinal Evaluation: You qualify for this arm of the study if you:
  1. Have a total hip replacement with a ceramic component
  2. Have a metal-on-polyethylene total hip replacement.
  3. Have your original or revised total hip replacement.
  You do not qualify for this arm of the study if you:
  1. Have occupational exposure to cobalt or chromium
  2. Have cemented components.
  3. Presence of a metal-on-metal (MOM) implant, or a recalled implant
  4. Standard contra-indications to MRI (e.g. cardiac pacemaker, etc.)

SUMMARY:
Patients with a total hip replacement may require early revision surgery due to an adverse local tissue reaction or bone resorption that occurs due to wear debris released from the implant. MRI provides a non-invasive biomarker for clinicians and surgeons to detect early adverse synovial reactions which may exist in the absence of clinical symptoms, thus imparting essential information for clinical management. This study will address two of the most commons causes of hip implant failure, including adverse local tissue reaction in implants not traditionally associated with adverse tissue reactions, as well as the presence of aseptic loosening and loss of implant-bone integration.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) has been successful in achieving pain reduction, but recent concerns have been raised regarding the development of adverse local tissue reactions (ALTRs). Our group has previously found that: 1) Magnetic resonance imaging (MRI) can detect and distinguish wear debris from THA; 2) MRI is sensitive to ALTR damage from different articulating surfaces; and 3) variable host-mediated response to wear debris mounts distinct morphologic patterns on MRI. There is continued interest in the evaluation of soft tissues near THAs as traditional THA designs, including metal-on-polyethylene (MOP) and ceramic-on-polyethylene (COP) bearing surfaces, have recently been implicated in ALTRs. It is believed that fretting and corrosion at the head-neck junction is responsible for ALTRs, secondary to flexural rigidity and other implant mechanical features. If a greater prevalence of ALTR is found in components with more flexible connections, this could drive the practice of THA to stiffer connections.

In this study, we will evaluate two important causes of implant failure: (1) in designs not traditionally associated with ALTRs such as metal-on-polyethylene (MOP) and ceramic-on-polyethylene (COP) we will assess patients indicated for revision THA surgery with MRI and correlate the imaging metrics to targeted biopsy retrieval obtained at the time of revision (including the trunnion), the extent of tissue damage documented at surgery, and implant retrieval analysis of the neck trunnion, including flexural rigidity analysis; and (2) to longitudinally assess implant integration using qualitative MRI evaluation of the bone-implant interface as well as quantitative MRI techniques, T2 mapping and T2* mapping using MAVRIC-UTE, to evaluate relaxometry at the interface.

ELIGIBILITY:
Inclusion Criteria:

Cohort #1:

1. Have a total hip replacement with a ceramic component undergoing revision for any reason, including recurrent dislocation.
2. Have a metal-on-polyethylene total hip replacement and have repeated dislocation, or
3. Have a metal-on-polyethylene total hip replacement greater than 1 year old, or
4. Have an infected total hip replacement (any surface bearing)

Cohort #2:

1. Have a total hip replacement with a ceramic component.
2. Have a metal-on-polyethylene total hip replacement.
3. Have your original or revised total hip replacement.

Exclusion Criteria:

Cohort #1:

1. Have occupational exposure to cobalt or chromium
2. Presence of MOM or recalled implant
3. Have had a prior revision of your total hip
4. Standard contra-indications to MRI

Cohort #2:

1. Have occupational exposure to cobalt or chromium.
2. Have cemented components.
3. Presence of a metal-on-metal or recalled implant.
4. Standard contra-indications to MRI.

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who will be having revision surgery of a total hip replacement, or individuals who currently have a total hip replacement with uncemented components.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Utilize MRI to evaluate total hip arthroplasty designs traditionally not implicated with the presence of adverse local tissue reactions. | An expected average of 1 year post-operatively
  All enrolled arthroplasty designs will be evaluated utilizing the input of:
  1. Evaluation of MR images: Presence, location, type and volume of synovitis, Synovial thickness, Impression of synovium, Presence and location of decompression of synovitis, Presence and location of low signal intensity deposits, Presence of soft tissue edema, Presence and location of dehiscence, Presence, location and volume of osteolysis, Assessment of implant loosening, Presence of and location of neurovascular compression, Disruption of abductors due to distended pseudocapsule, Presence of enlarged lymph nodes and presence and grading of adverse local tissue reaction.
  2. Pre-operative blood metal ion levels
  3. Pre-operative Hip disability and Osteoarthritis Outcome Score
  4. Pathologic evaluation of tissue obtained intra-operatively
  5. Intra-operative grade of soft tissues around the primary total hip replacement
  6. Implant wear analysis
Longitudinal monitor of arthroplasty loosening in patients with different individual risk factors and implant bearing surfaces and characteristics | This outcome will be measured at 4 different time points: Initial office visit, 1 year follow-up, 2 year follow-up, 3 year follow-up.
  All enrolled arthroplasty designs will be evaluated utilizing the input of:
  1. The formation a fibrous membrane and/or osteolysis around the implants
  2. Individual risk factors from subjects (gender, BMI, primary diagnosis, and level of activity)
  3. Individual risk factors based on implant characteristics (stem length, head size, and modular stem connections).

SECONDARY OUTCOMES:
Mode of total hip arthroplasty failure | An expected average of 1 year post-operatively
  Patients will be classified as symptomatic with mechanical symptoms and symptomatic with unexplained pain. These groups are based on the categories used by the National Joint Registry of England and Wales. Patients presenting with loosening, instability, or malalignment will be classified as "mechanical" failure. In cases of loosening, patients will be categorized as having acetabular or femoral loosening, only when documented intra-operatively by the surgeon. Patients presenting with pain not attributable to implant loosening, instability, or component malposition will be classified as "unexplained" failure. No specific unit of measure will be used for this outcome measure.
Blood serum metal ion levels | Measurement at an expected average of 1 year post operatively for revision total hip arthroplasty patients, or at initial office visit, 1 year follow-up, 2 year follow-up, and 3 year follow-up for individuals being monitored longitudinally.
  Blood samples will be drawn into lithium-heparin containing tubes with non-contamination precautions, and analyzed with high resolution inductively coupled mass spectrometry for the most accurate assessment of Cobalt and Chromium metal ion levels, to be measured in parts per million (ppm) or microgram per liter (ug/L)
Radiographic evaluation of implant orientation - anteversion and inclination | Measurement at an expected average of 1 year post operatively for revision total hip arthroplasty patients, or at initial office visit for individuals being monitored longitudinally.
  The assessment of hip replacement acetabular component position will be performed using the Einzel-Bild-Roentgen-Analysis (EBRA) software. The femoral stem-shaft angle will be measured in the frontal plane. The acetabular inclination angle will be measured in the frontal plane. The acetabular anteversion angle will be measured in the lateral plane. All measurements will be expressed in units of degrees.
MRI evaluation of soft tissues surrounding total hip arthroplasty | Measurement at an expected average of 1 year post operatively for revision total hip arthroplasty patients, or at initial office visit, 1 year follow-up, 2 year follow-up, and 3 year follow-up for individuals being monitored longitudinally.
  Evaluation of MR images: Presence, location, type and volume (measurement units of mm^3) of synovitis, Synovial thickness (measurement units of mm), Impression of synovium, Decompression of synovitis, Decompression into Trochanteric Bursa, Decompression into Iliopsoas, Presence and location of low signal intensity deposits, Presence of soft tissue edema, Presence and location of dehiscence, Presence, location and volume (measurement units of mm^3) of osteolysis, Assessment of implant loosening, Presence of and location of neurovascular compression, Disruption of abductors due to distended pseudocapsule, Presence of enlarged lymph nodes and presence and grading of adverse local tissue reaction. All quantitative values have the units of measurement indicated.
Intraoperative damage assessment | Measurement during revision surgery for total hip arthroplasty patients
  A subjective scoring system will be used for intraoperative damage assessment of the hip joint. The system is based on a 0 to 3 scale denoting the level of involvement of the soft tissues surrounding the joint (capsule, synovium, and muscle): 0 = Normal tissue; 1 = Fluid collection ± mild synovial reaction with or capsular dehiscence; 2 = the same findings as a score of 1, but with moderate synovial reaction; and 3 = the same findings as a score of 2, but with the addition of damage to the abductor muscle and/or osteolysis. No specific unit of measure will be used for this outcome measure.
Histologic analysis of retrieved tissues | Measurement at an expected average of 1 year post operatively for revision total hip arthroplasty patients.
  Histological evaluation will be using a 10 point aseptic lymphocytic vasculitis associated lesion (ALVAL) score to assess tissue reaction to a total hip replacement. The ALVAL score is a summation of individual grades assigned to the integrity of the synovial lining, presence and extent of inflammatory cell infiltrates, necrosis and tissue organization.
  We will use a supplemental grading system intended for metal-on-poly and ceramic implants since ALVAL grading is used primarily for metal-on-metal (MOM) articulations and may not detect similar features of wear debris in non-MOM articulations, polyethylene, metal or corrosion products. The presence of ceramic and polyethylene particles and the relative number of macrophages, giant cells, histiocytes, acute or chronic inflammatory cells, and presence of necrotic tissue will be graded using the scale of: 1) absent (-), little (+), moderate (++), extensive (+++). No specific unit of measure will be used for this outcome measure.
Implant retrieval wear analysis | Measurement at an expected average of 1 year post operatively for revision total hip arthroplasty patients.
  The bearing surfaces of the femoral heads and acetabular components, the neck trunnion of the total hip replacement femoral stems, and the matching female tapers of the total hip replacement heads retrieved at surgery will be scanned with a technique that utilizes a non-contact measurement method to calculate volumetric wear (measurement units of mm^3) and linear wear (measurement units of mm).
T2 Mapping of synovial tissues | Measurement at an expected average of 1 year post operatively for revision total hip arthroplasty patients.
  Quantitative imaging, specifically T2 mapping of soft tissues near the implant, specifically, the synovium and synovial volume.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew F Koff, PhD, Principal Investigator — Hospital for Special Surgery, New York; Hollis G Potter, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We will encourage the sharing of our final research data to enable further exploration of the data not presented in the application and for encouraging other individuals to develop new methods of data analysis. The data will be organized by subject number and by date of procedure (e.g. radiographs, MRI, serum metal ion levels, histology, wear analysis, etc.) for ease of identifying a specific dataset. The data will be stored on our servers and back-up drives. Individuals requesting electronic data will be given a link to a private web server to download the requested information, or will be requested to pay a nominal fee to burn the data to CD or DVD or to download to an individual's blank external hard drive, and for mailing charges depending on the type of data requested. Our goal is to make the data as easily accessible to the public as possible.
Supporting Information: Study Protocol
Time Frame: The data will become available within 1 year of study completion
Access Criteria: Data access requests will be reviewed by the primary investigators

REFERENCES:
- See also: Hospital for Special Surgery MRI Laboratory — http://www.hss.edu/research-magnetic-resonance-imaging-lab.asp

DOCUMENTS (1):
  • Informed Consent Form (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT02255331/ICF_000.pdf